CLINICAL TRIAL: NCT03178162
Title: Evaluation of a Non-invasive Cardiac Output Monitoring System in Comparison to the Semi-invasive Monitoring System FloTrac VigileoTechnology in Elderly Patients.
Brief Title: Evaluation of a Non-invasive Cardiac Output Monitoring System.
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Dr. Jochen Renner, PD Dr. Jochen Renner, University Hospital Schleswig-Holstein
Other Study IDs: IN-OCT-02
Record Dates: First submitted 2017-06-03; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Surgery in Elderly Patients; Hemodynamics; Pulse Wave Transit Time
Keywords: limitation in conventional monitoring

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are different methods for measuring cardiac output (CO) completely non-invasive, which are used today. Two of these should be used in the study to examine the CO in an older group of patients (> 65 years) undergoing major trauma surgery. The first method is the esCCOTM-technology by Nihon Kohden, the second uses the Volume Clamped Method via a finger-cuff by Nexfin Edwards life sciences. Both technologies work continuously and fully non-invasive.

The measured data will be compared to established standard procedures like semi-invasive pulse contour analysis using the Flotrac-Vigileo system. The study should answer the following questions:

How accurate and precise are the non-invasive methods? How large is the percentage deviation in comparison to the established standard? Are there any limitations of measuring accuracy regarding the age of the patient? The continuous hemodynamic monitoring of patients during surgery has recently changed from invasive and semi-invasive methods to completely non-invasive technologies. The accuracy and precision of this way of measuring cardiovascular parameters in comparison to the invasive standard is still controversial. Especially for older patient with atherosclerotic alteration of the blood vessels the utility of non-invasive monitoring systems is not shown yet. But principally this group with a high level of comorbidity might profit notably from less invasive procedures. This is the reason for the planed research.

DETAILED DESCRIPTION:
The Nexfin® monitoring system by Edwards life sciences could measure continuous non-invasive blood pressure through a finger-cuff for every single heart beat; moreover it calculates a CO and stroke-volume parameter utilizing a so-called pulse contour analysis provided by the non-invasive blood pressure measurement. This technology is based on an inflatable doublefinger-cuff wristband, which is attached to the patients hand and connected to a monitor. Using this wristband the arterial pressure within the patient's digital arteries will be continuously registered. Using a heart-frequency adapted algorithm - based on an alignment chart including healthy patients, patients with arterial hypertonia and micro/macro angiopathia - the software is also able to measure the brachial artery blood pressure.

First evaluations regarding non-invasive blood pressure measurement were very promising. However, data especially in elderly patients and patients with vascular disease are still not available.

The esCCO monitor (estimated Continuous Cardiac Output) by Nihon Kohden (Nihon Kohden Europe GmbH, 61191 Rosbach, Deutschland) is another completely non-invasive measurement device, which is based on the pulse wave transit time (PWTT) as well as non-invasive blood pressure measurement, ECG and pulse oximetry. PWTT provides time adapted information, e.g. intravascular pressure transmission or information on changes in the arterial blood volume.

Besides common vital signs such as SpO2, RR and ECG, esCCO™ also offers a realtime non-invasive CO-measurement. Mainly, the esCCO™ principle is based on the possibility to obtain CO-values using pulse pressure analysis: CO = SV × HR = (C × PP) × HR [SV: stroke volume; C: constant value; PP: Pulse Pressure; HR: Heart Rate]. Since studies have shown that there is a greater correlation between SV and PWTT than between SV and PP, the CO calculation was stated as followed as a result of the PWTT information: CO = SV × HR= C × (α × PWTT ＋ β) × HR = esCCO [α, β: experimental constants].

Demographic changes but also clinical everyday life indicates a strong increase in older patients undergoing surgery. The percentages of risk or high-risk patients with relevant comorbidities will therefore tremendously increase as well. If it is possible to adequately monitor this particular collective continuously with even less invasive technologies is to be answered by this clinical trial.

During surgery the hemodynamic parameters will be measured continuously and documented every 15 minutes or in special situation like hypotension or when vasoactive agents need to be given.

There will be no additional risk for the patient participating in the study, because the used devices and procedures have already been tested clinically. In general the preoperative preparation will be not different to the usual procedure. If a patient denies to participate the trial or withdraw his or her agreement afterwards there will be no disadvantage in terms of medical care for him or her. The people will be informed about this fact when he or she gives the agreement to the examination.

If a change of the surgical procedure or anaesthesia occurs its management will be given priority and the examination for the trial will stop quickly. Any adverse event potentially caused by the study will entail an interruption of the trial until its reason is found; the ethics committee will be informed immediately.

The planed clinical trial deals with the evaluation of different methods (invasive vs. non-invasive) to measure cardiac output and other parameters. For interpretation purpose the method of Bland and Altman will be used to calculate the average deviation (bias) and precesion (mean value ± 2 standard deviations). The mean percentage error will be determined in accordance to the criteria described by Critchley and Critchley. The Bland-Altman analysis will be expanded by repeated measurements per patient and point in time.

There is no mentionable, additional risk that the patient will be exposed to in course of the study since there is only monitoring systems being applied that are either fully clinically established or completely non-invasive.

Generated data will include common cardio-vascular parameters, such as: ECG, invasive as well as non-invasive blood pressure, oxygen saturation, endexpiratory CO2- partial pressure, cardiac output and stroke volume (both semi-invasively as well as non-invasively generated), echocardiographically generated data such as stroke volume, volume demand and cardiac output.

ELIGIBILITY:
Inclusion Criteria:

* Major surgery (elective or urgent) in vascular surgery and trauma surgery
* Patient´s rating according to ASA physical status classification system with 2-4
* Written consent by patient
* Age > 65

Exclusion Criteria:

* ASA 5
* Patient requiring high doses of catecholamine already before surgery
* Cognitive or language barriers restricting informant consent of patient
* Denial of participation by the patient
* emergency surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients older than 65 years who will participate in vascular or trauma surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
cardiac output | through study completion, an average of 1,5 years
  Comparison of cardiac output, utilizing cardiac index (CI), between (esCCO™ Nihon Khoden) and the Flotrac-Vigileo (Edward Lifesciences) monitoring system.

SECONDARY OUTCOMES:
pulse wave transit time (PWTT) | through study completion, an average of 1,5 years
  relevance of the measured time

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Schleswig-Holstein Campus Kiel - Klinik für Anästhesiologie und Operative Intensivmedizin, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No